CLINICAL TRIAL: NCT05128643
Title: Clinical Study on the Immunogenicity and Safety of the Recombinant Novel Coronavirus（COVID-19）Vaccine (CHO Cell) 0-1-6 Month and 0-1-4 Month Immunization Programs in People Aged 18 and Above
Brief Title: Clinical Study on the Immune Program of Recombinant Novel Coronavirus（COVID-19) Vaccine (CHO Cell)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIT-LKM-2021-NCV02
Record Dates: First submitted 2021-11-18; First posted 2021-11-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population Ⅰ (Experimental): At 0,1,6 months, 3 doses of experimental vaccine were injected into the deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant novel coronavirus vaccine (CHO cell)
- Population II (Experimental): At 0,1,4 months, 3 doses of experimental vaccine were injected into the deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant novel coronavirus vaccine (CHO cell)

INTERVENTIONS:
Biological: Recombinant novel coronavirus vaccine (CHO cell) — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose Recombinant novel coronavirus vaccine (CHO cells).

SUMMARY:
Popular topic：Clinical study on the immune program of recombinant Novel Coronavirus (COVID-19) vaccine (CHO cell). Research purpose:Main purpose: To evaluate the immunogenicity of recombinant novel coronavirus vaccine (CHO cells) inoculated at 0,1,6 months or 0,1,4 months in persons aged 18 years and over. Secondary purpose: To evaluate the safety of the investigational vaccine in people aged 18 and above.

Overall design: In this study, recombinant novel coronavirus vaccine (CHO cells) is inoculated at 0,1,6 months or 0,1,4 months in persons aged 18 years and older to evaluate the immunogenicity and safety.

Study population:The study involved people 18 years of age and older. Test groups：A total of 300 subjects were enrolled, including 221 in the 18-59 age group and 79 in the ≥60 age group. Three doses of experimental vaccine were administered according to the 0,1,6 month immunization schedule (Study No. 001-150) or 0,1,4 months immunization schedule (Study No. 151-300).

DETAILED DESCRIPTION:
Overall design:In this study, recombinant novel coronavirus vaccine (CHO cells) is inoculated at 0,1,6 months or 0,1,4 months in persons aged 18 years and older to evaluate the immunogenicity and safety.

Intervention: A total of 300 subjects were enrolled, including 221 in the 18-59 age group and 79 in the ≥60 age group. Three doses of experimental vaccine were administered according to the 0,1,6 month immunization schedule (Study No. 001-150) or 0,1,4 months immunization schedule (Study No. 151-300).

Immunogenicity observation:

About 5.0mL of venous blood was collected from all subjects for immunogenicity test before the first dose, before the third dose, on day 14 and 180 after full immunization.

Safety observation:

All adverse events (AE) were collected within 30 minutes after each dose, all AEs (both solicited and unsolicited) were collected 0-7 days after each dose, and all AEs (unsolicited) were collected 8-30 days after each dose. All SAEs were collected from the first dose up to 6 months after full immunization.

Solicited AEs (the following events occurring within 7 days of vaccination) :

Adverse events at the inoculation site (local) : pain, swelling, induration, redness, rash, pruritus; Vital signs: fever; Non-inoculated site (systemic) adverse events: headache, fatigue, diarrhea, nausea, vomiting, muscle pain (non-inoculated site), acute allergic reaction, cough.

Vital signs and physical examination:

1. All subjects underwent a daily armpit temperature examination during the screening period, before subsequent doses, and within 7 days after each dose.
2. All subjects underwent physical examination (skin and cardiopulmonary auscultation) and blood pressure measurement during the screening period.

ADE/VED (Antibody Enhancement/vaccine Enhancement disease) Risk Monitoring:

After vaccination (at least one dose of experimental vaccine), if the subject is diagnosed with COVID-19, he/she should go to the hospital for hospitalization or be isolated in accordance with the epidemic prevention and control requirements of the area in which he/she is located. A special investigation should be conducted for the existence of ADE/VED in severe/critical cases/deaths.

ELIGIBILITY:
Inclusion Criteria:

1. Persons over the age of 18 with full capacity for civil conduct;
2. The subject voluntarily agrees to participate in the study and signs the informed consent, and can provide valid identification, understand and comply with the requirements of the study protocol;
3. Fertile male and female subjects of reproductive age agreed to use effective contraceptive measures from the beginning of the study to 2 months after full vaccination.

Exclusion Criteria:

1. Suspected or confirmed fever within 72 hours before enrollment, or armpit temperature ≥37.3℃ on the day of enrollment;
2. Have a history of severe allergy to any component of the test vaccine, including aluminum preparation, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, dyspnea, angiopantic edema, etc.; Or have a history of severe adverse reactions to any of the above mentioned vaccines or medications;
3. people who currently have or have a history of COVID-19;
4. Persons suffering from the following diseases:

   ① have thrombocytopenia, any coagulation dysfunction or receive anticoagulant treatment, etc.;

   ② Congenital or acquired immune deficiency or autoimmune disease history or received immunomodulatory treatment within 6 months Treatment, such as immunosuppressive doses of glucocorticoid (dose reference: equivalent to prednisone 20mg/ day, more than one weeks); Or monoclonal antibodies; Or thymosin; Or interferon; However, topical application (e.g. ointments, eye drops) is allowed Liquid, inhalant or nasal spray);

   ③ Have been diagnosed with a known infectious disease, such as active tuberculosis, viral hepatitis, human immunodeficiency virus or treponema pallidum;

   ④ Neurological disorders (e.g., convulsions, migraines, epilepsy, stroke, epileptic seizures in the last three years, encephalopathy, focal neurological deficits, Guillain-Barre syndrome, encephalomyelitis or transverse myelitis); History of mental illness or family history;

   ⑤ functional absence of spleen, and absence of spleen or splenectomy caused by any reason;

   ⑥ There are serious chronic diseases or diseases in the progressive stage can not be controlled smoothly, such as diabetes, drugs can not control Hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg);

   ⑦ Severe liver and kidney diseases; Any current respiratory illness requiring routine medication (e.g., chronic obstructive pulmonary disease [COPD], asthma) or any exacerbation of respiratory illness (e.g., exacerbation of asthma) within the last 5 years; A history of serious cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease, arrhythmia, conduction block, myocardial infarction, pulmonary heart disease) or myocarditis or pericarditis;

   ⑧ Cancer patients (except basal cell carcinoma).
5. had taken an antipyretic or painkiller within 24 hours before the first dose of vaccine;
6. Those who have received novel coronavirus vaccine, or subunit vaccine and/or inactivated vaccine within 7 days before the first dose, or live attenuated vaccine within 14 days;
7. Have received blood or blood-related products, including immunoglobulin, within 3 months; Or planned for use during the study period;
8. Lactating or pregnant women (including women of childbearing age who have positive urine pregnancy test), or women who plan to have a pregnancy within 2 months after full vaccination of the test vaccine or their partners;
9. Have participated in or are currently participating in other COVID-19 related clinical trials;
10. The Investigator believes that the subject has any disease or condition that may place the subject at unacceptable risk; Subjects cannot meet the requirements of the program; Conditions that interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-04-12 (Estimated); Study Completion 2022-10-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity primary endpoint | 14 days after full immunization
  SARS-CoV-2 neutralizing antibody GMT

SECONDARY OUTCOMES:
Immunogenicity secondary endpoint | 14 days after full immunization
  positive conversion rate, positive rate, GMI of SARS-CoV-2 neutralizing antibody, RBD protein binding antibody (IgG); GMT of RBD protein binding antibody (IgG)
Immunogenicity secondary endpoint | 180 days after full immunization
  positive rate, GMT of SARS-CoV-2 neutralizing antibody, RBD protein binding antibody (IgG)
Safety endpoint | One month after each dose
  All adverse events (AEs)
Safety endpoint | From the first dose to 6 months after full immunization
  Incidence of all serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Huang Tao, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No